CLINICAL TRIAL: NCT04152187
Title: Investigation of the Effects of Inspiratory Muscle Training in Patients With Pulmonary Hypertension
Brief Title: Effects of Inspiratory Muscle Training in Patients With Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Buse Ozcan Kahraman, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pulmonary Hypertension; 2018.KB.SAG.099 (Other Grant/Funding Number: Dokuz Eylül University Scientific Research Coordination Unit)
Record Dates: First submitted 2019-11-02; First posted 2019-11-05 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Hypertension, Pulmonary
Keywords: pulmonary hypertension; inspiratory muscle training; muscle weakness
MeSH Terms: conditions — Hypertension, Pulmonary; Muscle Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training (IMT) (Experimental): Patients will receive IMT for 30 min (15x2), 7 times per week for 8 weeks using inspiratory muscle trainer device (PowerBreathe). During training, patients will be instructed to maintain diaphragmatic breathing. Inspiratory load will be set at 40-60% of maximum inspiratory pressure. Each week, six training sessions will be held at home and a training session will be supervised with physiotherapist.
  Interventions: Other: Inspiratory muscle training
- Control (No Intervention): No additional intervention

INTERVENTIONS:
Other: Inspiratory muscle training — The treatment group will receive inspiratory muscle training.
  Arms: Inspiratory muscle training (IMT)

SUMMARY:
This study aims to determine the possible effects of inspiratory muscle training on cardiovascular, respiratory, physical and psychosocial functions in patients with PH.

DETAILED DESCRIPTION:
Pulmonary Hypertension (PH) is a hemodynamic finding related to increase in pulmonary artery pressure. Because PH disease is a progressive, rare disease, it is important for this disease group to prolong the life span and to increase the quality of life and functional capacity. PH patients have been shown to have weakness in peripheral and respiratory muscles.

Patients will be randomly assigned to the inspiratory muscle training and control group. Inspiratory muscle training will be initiated in accordance with the patient at a range of 40-60%. İnspiratory muscle training will be given based on the assessments by the physiotherapist. Patients with PH who come to the routine outpatient clinic and volunteer will be included in the study. The first session will be the evaluation session and the 8-week inspiratory muscle training will be given, the other group will be the control group only. Dyspnoea, diaphragm thickness, pulmonary function, respiratory and peripheral muscle strength, blood pressure, arterial stiffness, physical activity, anxiety, depression and quality of life assessments will be repeated before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Pulmonary Hypertension
* According to the New York Heart Association functional class II - III
* Cases receiving stable medication for 3 months

Exclusion Criteria:

* Conditions which can limit the assessments
* Severe ischemic heart disease
* Acute cor pulmonale

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
6 minute walk test | Change from Baseline at 8 weeks
  functional capacity

SECONDARY OUTCOMES:
Mouth pressures | Change from Baseline at 8 weeks
  Maximal inspiratory pressure, maximal expiratory pressure and endurance will be measure with mouth pressure device
Modified Medical Research Council Dyspnea Scale | Change from Baseline at 8 weeks
  Modified Medical Research Council Dyspnea Scale is used to measure dyspnea. Higher scores indicate higher dyspnea.
Forced vital capacity | Change from Baseline at 8 weeks
  Forced vital capacity is defined as the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible.
Forced expiratory volume in 1 second | Change from Baseline at 8 weeks
  The volume of air expired in the first second of expiration or forced expiratory volume in 1 second, especially when expressed as a ratio with the total amount of air expired during the forced vital capacity, is a good index of expiratory airways resistance.
Diaphragma thickness | Change from Baseline at 8 weeks
  Diaphragma thickness will be measured by two dimensional ultrasonography
Levels of blood pressure | Change from Baseline at 8 weeks
  Ambulatory blood pressure monitoring will be used for blood pressure measurement
Arterial stiffness | Change from Baseline at 8 weeks
  During blood pressure measurements, augmentation index will be measured by non-invasive oscillations over the brachial artery.
Isometric muscle strength | Change from Baseline at 8 weeks
  Isometric muscle strength for knee extensors and shoulder flexors and abductors
Upper extremity exercise capacity | Change from Baseline at 8 weeks
  Upper extremity exercise capacity will be measured with Six-Minute Pegboard and Ring Test. In this test 4 iron rods, and a total of 20 rings are placed on a pegboard. At the end of six minutes, total number of rings placed will count.
International Physical Activity Questionnaire-Short Form | Change from Baseline at 8 weeks
  The International Physical Activity Questionnaire-Short Form has 7 items listing activities and requests estimates of durations and frequencies for each activity engaged in over the past week. Durations are multiplied by known metabolic equivalents per activity and the results for all items are summed for the overall physical activity score. Scores for walking and for moderate and vigorous activities are sums of corresponding item scores. Higher scores indicate higher physical activity level.
Fatigue Impact Scale | Change from Baseline at 8 weeks
  The Fatigue Impact Scale is widely used to measure fatigue. It is a 40-item multidimensional scale measuring the physical, cognitive and social. Patients are asked to rate how much of a problem fatigue has caused them during the past month, including the day of testing, on a 5-point Likert-type scale, with response options ranging from 0 "no problem" to 4 "extreme problem". Loer scores indicate the better results
Nottingham Health Profile | Change from Baseline at 8 weeks
  Health-related quality of life will be assessed using Nottingham Health Profile scale which is a general quality of life questionnaire that measures perceived health problems and their impact on normal daily activities. It has 38 items divided into six domains: energy level, pain, emotional reactions, sleep, social isolation and physical abilities. Items use yes/no answer format and each item is weighted. Total scores for each domain range from 0 to 100. Higher scores represent less quality of life in relevant domain.
Changes in Anxiety and Depression | Change from Baseline at 8 weeks
  Anxiety and depression levels will be assessed by Hospital Anxiety and Depression Scale. The scale consists of 14 items, seven items for the anxiety subscale and seven for the depression subscale. Each item is scored on a response-scale with four alternatives ranging between 0 and 3. Higher scores indicate
Changes in Dyspnea | Change from Baseline at 8 weeks
  Dyspnea level will be questioned with the modified Borg Scale. Minimum value is 0 (no dyspnea), and maximum value is 10 (maximal dyspnea) Higher scores indicate higher fatigue levels.

CONTACTS AND LOCATIONS:
Overall Officials: Buse Ozcan Kahraman, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylül University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No